CLINICAL TRIAL: NCT02169050
Title: Vitamin D, Inflammation, and Relations to Insulin Resistance in Morbidly Obese Pre-Menopausal Women
Brief Title: Association Between Vitamin D and Inflammation and Diabetes Risk in Morbidly Obese Pre-Menopausal Women
Acronym: VitD2014
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-1010
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Insulin Sensitivity
Keywords: Vitamin D deficiency; Inflammation; Obesity
MeSH Terms: conditions — Insulin Resistance; Vitamin D Deficiency; Inflammation; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Plasma Adipose tissues
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No intervention: There is no intervention to subjects in this study. All subjects are morbidly women seeking bariatric surgeries.

SUMMARY:
Obesity is associated with low-grade inflammation, insulin resistance and low vitamin D status. Vitamin D has traditionally been known to involve in calcium homeostasis and prevent rickets; however, recently it has been recognized to inversely associate with many non-skeletal diseases and conditions including obesity and type 2 diabetes (T2DM). In vitro studies have demonstrated that vitamin D possesses anti-inflammatory properties. It remains unknown if the effect of vitamin D on insulin sensitivity is mediated by suppressing inflammation in human adipose tissues. The main objective of this study was to assess the association between vitamin D and insulin sensitivity and inflammation in morbidly obese pre-menopausal women. Obese women (n=76) were recruited from the University of Illinois at Chicago (UIC) Nutrition and Wellness Center and the UIC medical center bariatric surgery clinics. Insulin sensitivity/resistance was assessed by (1) Oral glucose insulin sensitivity (OGIS) index, derived from dynamic oral glucose tolerance test (OGTT), and (2) Homeostasis model of insulin resistance (HOMA-IR), calculated from fasting steady-state glucose and insulin. Also, to better understand the potential mechanism and the role circulating vitamin D (25OHD) plays in adipose tissue inflammation, we assessed messenger ribonucleic acid (mRNA) expression of vitamin D receptor (VDR) and various inflammatory genes in visceral (VAT) and subcutaneous adipose tissues (SAT) of obese women that underwent a restrictive bariatric procedure. We hypothesized that subjects with higher serum vitamin D levels would be less inflamed and more insulin sensitive and have increased expression of VDR and pro-inflammatory markers compared to those with lower serum vitamin D levels.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between the age of 21 and 49 years old
* BMI >=35(kg/m2)
* Not pregnant
* English speaking
* Approved for a bariatric surgery

Exclusion Criteria:

Subjects with:

* Diabetes
* Cancer
* Kidney disease
* Liver disease
* Gallbladder disease
* Rheumatoid arthritis
* HIV/AIDS
* Crohn's disease or inflammatory bowel disease
* Subjects taking anti-inflammatory medications

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study subjects are drawn from women seeking surgical treatment for their morbid obesity at the University of Illinois at Chicago Medical Center (UICMC) Bariatric surgery clinics.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2011-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Oral Glucose Insulin Sensitivity (OGIS) | 2 hour, 1-5 weeks before bariatric surgery
  Insulin sensitivity is assessed based with a 2-hour, 75gm Oral Glucose Tolerance Test. Blood samples are collected at 0, 90, and 120 min for the measurement of glucose and insulin.

SECONDARY OUTCOMES:
Adipose tissue mRNA Expression of Vitamin D Receptors and Inflammation Markers | 10-20 minutes, during bariatric surgery
Inflammatory markers in plasma | 3-15 minutes, 1-5 weeks before bariatric surgery
  Fasting blood drawn on Oral Glucose Tolerance Test day, which is 1-5 weeks before bariatric surgeries

CONTACTS AND LOCATIONS:
Overall Officials: Carol Braunschweig, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States